CLINICAL TRIAL: NCT01714492
Title: In Vivo Mechanics Analysis of Patients Having a Sigma Mobile Bearing TKA
Brief Title: Mechanics Analysis of Patients Having a Sigma Mobile Bearing TKA
Acronym: Sigma MB TKA
Status: Completed | Type: Observational
Sponsor: The University of Tennessee, Knoxville (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Principal Investigator, Richard Komistek, Principal Investigator, The University of Tennessee, Knoxville
Other Study IDs: 11019; R01 1373 424 (Other: The University of Tennessee)
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Results first posted 2014-02-17 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2019-10

CONDITIONS: Knee Prosthesis; Knee Replacement Arthroplasty
Keywords: Total Knee Arthroplasty (TKA); in vivo mechanics; kinematics; fluoroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly: subjects implanted with the Sigma Posterior Stabilizing Rotating Platform TKA including a polyethylene insert with 4 beads
  Interventions: Device: Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly

INTERVENTIONS:
Device: Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly — Sigma PS RP TKA including a polyethylene insert with 4 beads

SUMMARY:
Utilize previously developed mathematical model to determine in vivo knee mechanics (kinematics, forces, stresses, areas and sound) for subjects having a Sigma Posterior Stabilizing (PS) mobile bearing (MB) total knee arthroplasty (TKA). There are several hypotheses for this study, although the most prominent is: Subjects having a Sigma RP PS TKA will experience polyethylene bearing rotation at 10 years post-operative, similar to their previous evaluations at six months, two years and five years.

DETAILED DESCRIPTION:
Additional hypotheses:

* Subjects having a Sigma RP PS TKA will experience full ideal femorotibial contact mechanics.
* Subjects having a Sigma RP PS TKA will experience optimal cam/post mechanics.
* Subjects having a Sigma RP PS TKA will experience continuous axial rotation in deep flexion.
* Subjects having a Sigma RP PS TKA will experience optimal distribution of tibio-femoral and cam/post contact forces over a broad area on the post.
* Subjects having a Sigma RP PS TKA will experience a smooth transition of the cam on the post, not an abrupt slide as seen with fixed bearing PS TKA.
* The use of the sound sensors will detect cam/post contact mechanics under in vivo conditions.

ELIGIBILITY:
Inclusion Criteria:

* At least six months post-operative
* Between 40-85 years of age
* Have a body weight of less than 250 lbs.
* Judged clinically successful with a AKS greater than 90
* Have the DePuy Sigma mobile bearing TKA
* Good-to-excellent post-operative passive flexion
* Must be willing to sign the IC and HIPAA forms.

Exclusion Criteria:

* Pregnant females
* Those not willing to sign the IC and HIPAA forms

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are eight mobile bearing subjects that were implanted over 10 years ago with a custom polyethylene insert that has four beads rigidly inserted into the polyethylene component.
Sampling Method: Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2012-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard D Komistek, Ph. D., Principal Investigator — The University of Tennessee; Dennis A Douglas, MD, Principal Investigator — Colorado Joint Replacement
Locations (3):
- United States (3):
  - Porter Adventist Hospital, Colorado Joint Replacement, Denver, Colorado
  - Perkins Hall, The University of Tennessee, Knoxville, Tennessee
  - Science and Engineering Research Facility, The University of Tennessee, Knoxville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: hospital, medical clinic
Groups:
- Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly: subjects implanted with the Sigma Posterior Stabilizing Rotating Platform TKA including a polyethylene insert with 4 beads that allow for determination of polyethylene rotation.
Period: Overall Study
Arm/Group | Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 74 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 8

OUTCOME MEASURES:

1. Primary Outcome: In Vivo Linear Knee Kinematics From Fluoroscopy Evaluation During Deep Knee Bend Activity
Description: The values that were reported indicate the motion of the contact point from full extension to patient's maximum flexion. Throughout flexion, if the point translated forward (anteriorly) atop the tibial tray, the number was reported as positive. If the point traveled backwards (posteriorly) atop the tibial tray, the number was reported as negative.
Time Frame: 10 yrs post-operative
Population: Subjects implanted with the Sigma Posterior Stabilizing Rotating Platform TKA including a polyethylene insert with 4 beads that allow for determination of polyethylene rotation.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Implants
Groups:
- In Vivo Knee Kinematics From Fluoroscopy Evaluation During Dee: subjects implanted with the Sigma Posterior Stabilizing Rotating Platform TKA including a polyethylene insert with 4 beads that allow for determination of polyethylene rotation.
Arm/Group | In Vivo Knee Kinematics From Fluoroscopy Evaluation During Dee
Number analyzed (Participants) | 8
Number analyzed (Implants) | 8
mm
  Lateral Anterior Posterior Deep Knee Bend | -4.1 (2.4)
  Medial Anterior Posterior Deep Knee Bend | 1.2 (2.8)

2. Secondary Outcome: In Vivo Knee Force Values From Fluoroscopy Evaluation During Deep Knee Bend Activity
Description: The intended unit of measure is "times Body Weight" (or xBW), relating to a ratio.
Time Frame: 10 yrs post-operative
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: times body weight
Units Other Than Participants: Implants
Arm/Group | Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly
Number analyzed (Participants) | 8
Number analyzed (Implants) | 8
times body weight
  Medial Condyle Knee Force at Maximum Flexion | 1.57 (0.53)
  Lateral Condyle Knee Force at Maximum Flexion | 1.39 (0.36)

3. Primary Outcome: Femoral Axial Rotation With Respect to the Tibia During Deep Knee Bend Activity
Time Frame: 10 yrs post-operative
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Implants
Arm/Group | In Vivo Knee Kinematics From Fluoroscopy Evaluation During Dee
Number analyzed (Participants) | 8
Number analyzed (Implants) | 8
degrees | 6.1 (5.8)

4. Primary Outcome: Range of Motion During Flexion of Deep Knee Bend Activity
Time Frame: 10 yrs post-operative
Measure: Mean (Standard Deviation); unit: degrees
Units Other Than Participants: Implants
Arm/Group | In Vivo Knee Kinematics From Fluoroscopy Evaluation During Dee
Number analyzed (Participants) | 8
Number analyzed (Implants) | 8
degrees | 103 (11.2)

5. Secondary Outcome: Condyle Contact Area at Maximum Flexion During Deep Knee Bend Activity
Time Frame: 10 yrs post-operative
Measure: Mean (Standard Deviation); unit: mm^2
Units Other Than Participants: Implants
Arm/Group | In Vivo Knee Kinematics From Fluoroscopy Evaluation During Dee
Number analyzed (Participants) | 8
Number analyzed (Implants) | 8
mm^2
  Medial | 109.16 (2.82)
  Lateral | 104.78 (21.22)

6. Secondary Outcome: Condyle Contact Stress at Maximum Flexion During Deep Knee Bend Activity
Time Frame: 10 yrs post-operative
Measure: Mean (Standard Deviation); unit: MPa
Units Other Than Participants: Implants
Arm/Group | In Vivo Knee Kinematics From Fluoroscopy Evaluation During Dee
Number analyzed (Participants) | 8
Number analyzed (Implants) | 8
MPa
  Average Medial Condyle Contact Stress | 10.66 (1.75)
  Average Lateral Condyle Contact Stress | 10.05 (1.45)

ADVERSE EVENTS:
Description: There were no adverse effects or events encountered for any subjects for this study.
Arm/Group | Sigma Posterior Stabilizing Rotating Platform TKA Beaded Poly
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Small study population; only one specific type of mobile bearing implant was analyzed; no definitive way to quantitatively measure level of wear on various implants to determine if there was any influence on the kinematic performance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes